CLINICAL TRIAL: NCT03242395
Title: Perioperative Research Into Memory (PRiMe): The Use of fMRI to Investigate Neuroinflammation, Cognitive Dysfunction and Quality of Life Following a Major Burn Injury and Critical Care Admission
Brief Title: PRIME: Cognitive Outcome Following Major Burns
Acronym: PRIME
Status: Completed | Type: Observational
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: University of Westminster (Other); Imperial College Healthcare NHS Trust (Other); Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 14/LO/0049
Record Dates: First submitted 2017-04-21; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2016-12

CONDITIONS: Cognitive Dysfunction; Burns; Inflammation, Brain; Quality of Life; Anxiety; Depression; PostTraumatic Stress Disorder
Keywords: Neuroinflammation; fMRI; Post-operative cognitive dysfunction; Systemic inflammation; Severe burns
MeSH Terms: conditions — Cognitive Dysfunction; Burns; Encephalitis; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Burn patients: Adult survivors of severe burns who have been admitted to Burns ITU for invasive ventilation within 10 years of neurocognitive assessment
- Controls: Healthy volunteers, controlled for age/sex/IQ

SUMMARY:
PRIME aims to demonstrate through neurocognitive assessment that BICU patients will have a degree of neurocognitive dysfunction following a major burn, that this neurocognitive dysfunction is due to an underlying neuroinflammatory process by fMRI neuroimaging techniques, and that the neurocognitive deficit is associated with a reduced quality of life.

DETAILED DESCRIPTION:
Patients were matched with for age, sex and IQ (as determined by National Adult Reading Test scores) controlled volunteers.

Participants were assessed for the following domains: verbal ability, verbal and visual learning, short-term memory, working memory, executive function, attention and processing speed. The domains were assessed with the following validated cognitive tests: The Hopkins Verbal Learning Test, Trail making parts A and B, phonemic, semantic and switching verbal fluency as well as the Cogstate computerised battery: Identification speed, Detection speed, One Card Learning accuracy, One Back test accuracy, Two Back test accuracy, International Shopping List total correct answers and Groton Maze Learning total errors. Evidence of neuroinflammation was assessed using an fMRI protocol (Resting state MRI, T1w-MPR, T2 Space, Diffusion Tensor Imaging with 30 directions, right frontal white matter and posterior cingulate gyrus Single Voxel Spectroscopy, and patient group Susceptibility Weighted Imaging.

Quality of life was measured using the EuroQoL 5 Dimensions and visual analogue scale. Independent Activities of Daily Living was also assessed. Mental Health (as a confounder) was measured using the Patient Health Questionnaire 9, the Beck Depression Index II, the Beck Anxiety Inventory and the Trauma Screening Questionnaire.

Statistical methods include significant differences between the patient and control group using the Student t test (parametric data), the Mann Witney U test (non parametric data) or the Fisher's Exact test (qualitative scoring systems). MELODIC in FSL software was used to decompose the rs-fMRI data into brain networks using independent component analysis (ICA) and connectivity in these networks patients and controls was compared using dual regression. FreeSurfer was used to extract brain regions from T1 images and compare the normalised volume of the hippocampus, amygdala and precuneus for patients and controls. DTI data were analysed using tract based spatial statistics (TBSS) in FSL and using FreeSurfer regions for the hippocampus, amygdala and precuneus. Cho/Cr, Cho/NAA and Ins/Cr ratios were extracted from MRS data using Tarquin. SWI images were reviewed for the presence of microbleeds by two Radiologists.

ELIGIBILITY:
Inclusion Criteria:

* Invasive ventilation on a Burns Intensive Care Unit (BICU) within the previous ten years
* Burn injuries greater than 15% total body surface area (TBSA)
* Adult

Exclusion Criteria:

* Admission to BICU for other illnesses that were not burn related (such as Toxic Epidermal Necrolysis Syndrome)
* Evidence of head trauma
* Known substance misuse or alcohol excess
* Inability to understand plain verbal or written English
* Severe mental health issues
* Receiving formal psychiatric treatment
* Currently held under the Mental Health Act
* If the subject's psychological health was deemed to be at risk from inclusion
* Imprisoned
* Contraindications to MRI
* non-compatible pacemakers
* surgical metalwork or foreign bodies
* severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Severe burns survivors
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Neurocognitive deficit | Within 10 years of injury
  Median T score of cognitive results (verbal ability, verbal and visual learning, short-term memory, working memory, executive function, attention and processing speed)

SECONDARY OUTCOMES:
Quality of Life | Within 10 years of injury
  EuroQoL 5D score
Neuroinflammation | Within 10 years of injury
  As per the functional Magnetic Resonance Imaging protocol

CONTACTS AND LOCATIONS:
Overall Officials: Marcela P Vizcaychipi, MD PhD, Principal Investigator — Anaesthetic and Intensive Care Consultant
Locations (1):
- Chelsea and Westminster Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No